CLINICAL TRIAL: NCT01241552
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Adaptive Design Study of the Efficacy, Safety, and Tolerability of a Single Infusion of MK-3415 (Human Monoclonal Antibody to Clostridium Difficile Toxin A), MK-6072 (Human Monoclonal Antibody to Clostridium Difficile Toxin B), and MK-3415A (Human Monoclonal Antibodies to Clostridium Difficile Toxin A and Toxin B) in Patients Receiving Antibiotic Therapy for Clostridium Difficile Infection (MODIFY I)
Brief Title: A Study of MK-3415, MK-6072, and MK-3415A in Participants Receiving Antibiotic Therapy for Clostridium Difficile Infection (MK-3415A-001)
Acronym: MODIFY I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3415A-001
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; recurrent Clostridium difficile; vancomycin; metronidazole; monoclonal antibody; Clostridium difficile infection (CDI)
MeSH Terms: conditions — Clostridium Infections | interventions — actoxumab; bezlotoxumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MK-3415 + SOC (Experimental): Single intravenous (IV) infusion of 10 mg/kg MK-3415 + Standard of Care for CDI
  Interventions: Biological: MK-3415; Drug: SOC
- MK-6072 + SOC (Experimental): Single IV infusion of 10 mg/kg MK-6072 + Standard of Care for CDI
  Interventions: Biological: MK-6072; Drug: SOC
- MK-3415A + SOC (Experimental): Single IV infusion of 10 mg/kg MK-3415A + Standard of Care for CDI
  Interventions: Biological: MK-3415A; Drug: SOC
- Placebo + SOC (Placebo Comparator): Normal saline infusion (0.9% sodium chloride) + Standard of Care for CDI
  Interventions: Biological: Placebo; Drug: SOC

INTERVENTIONS:
Biological: MK-3415 — A single IV infusion of MK-3415 (10 mg/kg of monoclonal antibody to Clostridium difficile Toxin A)
  Arms: MK-3415 + SOC
Biological: MK-6072 — A single infusion of MK-6072 (10 mg/kg of monoclonal antibody to Clostridium difficile Toxin B)
  Arms: MK-6072 + SOC
Biological: MK-3415A — A single IV infusion of MK-3415A (10 mg/kg of monoclonal antibody to Clostridium difficile Toxin A and 10mg/kg of monoclonal antibody to Clostridium difficile Toxin B)
  Arms: MK-3415A + SOC
Biological: Placebo — A single IV infusion of normal saline (0.9% sodium chloride)
  Arms: Placebo + SOC
Drug: SOC — Standard of care (SOC) for CDI will be prescribed for 10 to 14 days and can begin on the day of study drug infusion; but the first dose must have been administered prior to or within a few hours following study drug infusion. SOC is defined as the receipt of oral metranidazole, oral vancomycin, IV metronidazole concurrent with oral vancomycin, oral fidaxomicin, or oral fidaxomicin concurrent with IV metronidazole.

SUMMARY:
This study will investigate whether: 1) treatment with MK-3415A in addition to standard of care (SOC) antibiotic therapy will decrease Clostridium difficile infection (CDI) recurrence as compared to treatment with MK-6072 or MK-3415, 2) treatment with MK-3415A, MK-6072, or MK-3415, in addition to SOC antibiotic therapy will decrease CDI recurrence as compared to placebo, and 3) MK-3415A, MK-6072, and MK-3415 will be generally well tolerated in participants receiving SOC therapy for CDI as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* participant has a confirmed diagnosis of CDI as defined by: a. diarrhea, as defined by passage of 3 or more loose stools in 24 or fewer hours, AND b. A positive test for toxigenic C. difficile from a stool collected no more than 7 days before study infusion.
* participant must be receiving SOC therapy for CDI. SOC therapy is defined as the receipt of oral metronidazole, oral vancomycin, IV metronidazole concurrent with oral vancomycin, oral fidaxomicin, or oral fidaxomicin concurrent with IV metronidazole.
* participant is highly unlikely to become pregnant or to impregnate a partner since they meet at least one of the following criteria: a. A female participant who is not of reproductive potential is eligible without requiring the use of contraception. A female participant who is not of reproductive potential is defined as: one who has either (1) reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels in the postmenopausal range as determined by the local laboratory, or 12 months of spontaneous amenorrhea); (2) 6 weeks post surgical bilateral oophorectomy with or without hysterectomy; or (3) bilateral tubal ligation. Spontaneous amenorrhea does not include cases for which there is an underlying disease that causes amenorrhea (e.g. anorexia nervosa). b. A participant who is of reproductive potential agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control starting at enrollment and through the 12 Week study period. Acceptable methods of birth control are: intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, vasectomy and any registered and marketed hormonal contraceptives that contain an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents)
* participant or legal representative must have voluntarily agreed to participate by providing written informed consent after the nature of the study has been fully explained.

Exclusion Criteria:

* participant with an uncontrolled chronic diarrheal illness such that their normal 24-hour bowel movement habit is 3 or more loose stools.
* participant with a planned surgery for CDI within 24 hours.
* participant has a positive pregnancy test in the 48 hours before the infusion or is unwilling to undergo pregnancy testing if a pre-menopausal female who is not sterilized and therefore has the potential to bear a child.
* participant is breast-feeding or plans to breast-feed prior to the completion of the 12-week study period.
* A female participant who plans to donate ova prior to the completion of the 12-week study period, or a male participant who is planning to impregnate or provide sperm donation prior to the completion of the 12-week study period.
* participant has previously participated in this study, has previously received MK-3415 or MK- 6072 (either alone or in combination), has received a C. difficile vaccine, or has received another experimental monoclonal antibody against C. difficile toxin A or B.
* participant plans to donate blood and/or blood products within 6 months following the infusion.
* participant has received immune globulin within 6 months prior to receipt of the infusion or is planning to receive immune globulin prior to the completion of the 12-week study period.
* treatment with SOC therapy is planned for longer than 14 days.
* participant has received more than a 24-hour regimen of cholestyramine, colestimide, rifaximin, or nitazoxanide within 14 days prior to receipt of the infusion or is planning to receive these medications prior to the completion of the 12-week study period.
* participant plans to take medications that are given to decrease gastrointestinal peristalsis, such as loperamide (Imodium™) or diphenoxylate hydrochloride/atropine sulfate (LOMOTIL™), at any time during the 14 days following infusion. Participants receiving opioid medications at the onset of diarrhea may be included if they are on a stable dose or if there is anticipation of a dose decrease or cessation of use.
* participant plans to take the probiotic Saccharomyces boulardii or receive fecal transplant therapy, or any other therapies that have been demonstrated to decrease CDI recurrences at any time following infusion (Day 1) and through the completion of the 12-week study period.
* participant has received another investigational study agent within the previous 30 days, or is currently participating in or scheduled to participate in any other clinical trial with an investigational agent during the 12-week study period.
* participant is not expected to survive for 72 hours.
* participant has any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the participant participating in the study, would make it unlikely for the participant to complete the study, or would confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2014-12-09 (Actual); Study Completion 2014-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Zhang H, Mehrotra DV, Shen J. AWOT and CWOT for genotype and genotype-by-treatment interaction joint analysis in pharmacogenetics GWAS. Bioinformatics. 2023 Jan 1;39(1):btac834. doi: 10.1093/bioinformatics/btac834. PMID 36661328
- [Derived] Bouza E, Cornely OA, Ramos-Martinez A, Plesniak R, Ellison MC, Hanson ME, Dorr MB. Analysis of C. difficile infection-related outcomes in European participants in the bezlotoxumab MODIFY I and II trials. Eur J Clin Microbiol Infect Dis. 2020 Oct;39(10):1933-1939. doi: 10.1007/s10096-020-03935-3. Epub 2020 Jun 6. PMID 32504314
- [Derived] Shen J, Mehrotra DV, Dorr MB, Zeng Z, Li J, Xu X, Nickle D, Holzinger ER, Chhibber A, Wilcox MH, Blanchard RL, Shaw PM. Genetic Association Reveals Protection against Recurrence of Clostridium difficile Infection with Bezlotoxumab Treatment. mSphere. 2020 May 6;5(3):e00232-20. doi: 10.1128/mSphere.00232-20. PMID 32376702
- [Derived] Cornely OA, Mullane KM, Birch T, Hazan-Steinberg S, Nathan R, Bouza E, Calfee DP, Ellison MC, Wong MT, Dorr MB. Exploratory Evaluation of Bezlotoxumab on Outcomes Associated With Clostridioides difficile Infection in MODIFY I/II Participants With Cancer. Open Forum Infect Dis. 2020 Jan 31;7(2):ofaa038. doi: 10.1093/ofid/ofaa038. eCollection 2020 Feb. PMID 32099847
- [Derived] Kelly CP, Poxton IR, Shen J, Wilcox MH, Gerding DN, Zhao X, Laterza OF, Railkar R, Guris D, Dorr MB. Effect of Endogenous Clostridioides difficile Toxin Antibodies on Recurrence of C. difficile Infection. Clin Infect Dis. 2020 Jun 24;71(1):81-86. doi: 10.1093/cid/ciz809. PMID 31628838
- [Derived] Montgomery DL, Matthews RP, Yee KL, Tobias LM, Dorr MB, Wrishko RE. Assessment of Bezlotoxumab Immunogenicity. Clin Pharmacol Drug Dev. 2020 Apr;9(3):330-340. doi: 10.1002/cpdd.729. Epub 2019 Aug 14. PMID 31411386
- [Derived] Basu A, Prabhu VS, Dorr MB, Golan Y, Dubberke ER, Cornely OA, Heimann SM, Pedley A, Xu R, Hanson ME, Marcella S. Bezlotoxumab Is Associated With a Reduction in Cumulative Inpatient-Days: Analysis of the Hospitalization Data From the MODIFY I and II Clinical Trials. Open Forum Infect Dis. 2018 Nov 15;5(11):ofy218. doi: 10.1093/ofid/ofy218. eCollection 2018 Nov. PMID 30460321
- [Derived] Yee KL, Kleijn HJ, Kerbusch T, Matthews RP, Dorr MB, Garey KW, Wrishko RE. Population Pharmacokinetics and Pharmacodynamics of Bezlotoxumab in Adults with Primary and Recurrent Clostridium difficile Infection. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01971-18. doi: 10.1128/AAC.01971-18. Print 2019 Feb. PMID 30455246
- [Derived] Kelly CP, Wilcox MH, Glerup H, Aboo N, Ellison MC, Eves K, Dorr MB. Bezlotoxumab for Clostridium difficile Infection Complicating Inflammatory Bowel Disease. Gastroenterology. 2018 Oct;155(4):1270-1271. doi: 10.1053/j.gastro.2018.06.080. Epub 2018 Sep 15. No abstract available. PMID 30227108
- [Derived] Prabhu VS, Cornely OA, Golan Y, Dubberke ER, Heimann SM, Hanson ME, Liao J, Pedley A, Dorr MB, Marcella S. Thirty-Day Readmissions in Hospitalized Patients Who Received Bezlotoxumab With Antibacterial Drug Treatment for Clostridium difficile Infection. Clin Infect Dis. 2017 Oct 1;65(7):1218-1221. doi: 10.1093/cid/cix523. PMID 30060024
- [Derived] Birch T, Golan Y, Rizzardini G, Jensen E, Gabryelski L, Guris D, Dorr MB. Efficacy of bezlotoxumab based on timing of administration relative to start of antibacterial therapy for Clostridium difficile infection. J Antimicrob Chemother. 2018 Sep 1;73(9):2524-2528. doi: 10.1093/jac/dky182. PMID 29788418
- [Derived] Gerding DN, Kelly CP, Rahav G, Lee C, Dubberke ER, Kumar PN, Yacyshyn B, Kao D, Eves K, Ellison MC, Hanson ME, Guris D, Dorr MB. Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection in Patients at Increased Risk for Recurrence. Clin Infect Dis. 2018 Aug 16;67(5):649-656. doi: 10.1093/cid/ciy171. PMID 29538686
- [Derived] Wilcox MH, Gerding DN, Poxton IR, Kelly C, Nathan R, Birch T, Cornely OA, Rahav G, Bouza E, Lee C, Jenkin G, Jensen W, Kim YS, Yoshida J, Gabryelski L, Pedley A, Eves K, Tipping R, Guris D, Kartsonis N, Dorr MB; MODIFY I and MODIFY II Investigators. Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection. N Engl J Med. 2017 Jan 26;376(4):305-317. doi: 10.1056/NEJMoa1602615. PMID 28121498
- [Derived] Desai K, Gupta SB, Dubberke ER, Prabhu VS, Browne C, Mast TC. Epidemiological and economic burden of Clostridium difficile in the United States: estimates from a modeling approach. BMC Infect Dis. 2016 Jun 18;16:303. doi: 10.1186/s12879-016-1610-3. PMID 27316794

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants 18 years of age or older, with a diagnosis of Clostridium difficile Infection (CDI) were enrolled in this trial.
Groups:
- MK-3415 + SOC: Single intravenous (IV) infusion of 10 mg/kg MK-3415 + Standard of Care (SOC) for CDI
Period: Overall Study
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Started | 242 | 403 | 403 | 404
Treated | 235 | 392 | 388 | 397
Completed | 201 | 340 | 343 | 340
Not Completed | 41 | 63 | 60 | 64
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Death | 26 | 30 | 20 | 25
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Technical Problems | 2 | 0 | 2 | 2
Not completed — Progressive Disease | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 2 | 6 | 1
Not completed — Withdrawal by Subject | 7 | 15 | 14 | 15
Not completed — Physician Decision | 2 | 4 | 2 | 3
Not completed — Lost to Follow-up | 2 | 11 | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 242 | 403 | 403 | 404 | 1452
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (16.8) | 61.1 (18.5) | 62.5 (17.8) | 62.9 (18.3) | 62.5 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 238 | 224 | 230 | 829
  Male | 105 | 165 | 179 | 174 | 623

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clostridium Difficile Infection (CDI) Recurrence
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive local or central lab stool test for toxigenic Clostridium (C.) difficile following clinical cure of the initial CDI episode
Time Frame: Up to 12 weeks
Population: Participants who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 232 | 386 | 383 | 395
Percentage of participants | 25.9 | 17.4 | 15.9 | 27.6
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.3182, Miettinen and Nurminen — One sided p-value based on the Miettinen and Nurminen method stratified by SOC therapy (metronidazole vs. vancomycin vs. fidaxomicin) and hospitalization status (inpatient vs. outpatient); Adjusted Difference = -1.7, 95% CI 2-sided [-8.6 to 5.5] — Adjusted Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0003, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -10.1, 95% CI 2-sided [-15.9 to -4.3] — Adjusted Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -11.6, 95% CI 2-sided [-17.4 to -5.9] — Adjusted Difference: MK-3415A + SOC - Placebo + SOC
Statistical Analysis 4: Comparison: MK-3415 + SOC vs MK-3415A + SOC; Test type: Superiority or Other; p = 0.0013, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -9.9, 95% CI 2-sided [-16.9 to -3.4] — Adjusted Difference: MK-3415A + SOC - MK-3415 + SOC
Statistical Analysis 5: Comparison: MK-6072 + SOC vs MK-3415A + SOC; Test type: Superiority or Other; p = 0.2997, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -1.4, 95% CI 2-sided [-6.7 to 3.9] — Adjusted Difference: MK-3415A + SOC - MK-6072 + SOC

2. Secondary Outcome: Percentage of Participants With Global Cure
Description: Global Cure is defined as the clinical cure of the initial CDI episode and no CDI recurrence through Week 12. Clinical cure is defined as participants who received ≤ 14 day regimen of SOC therapy and have no diarrhea (≤2 loose stools per 24 hours) for two consecutive days following completion of SOC therapy for the initial CDI episode.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 232 | 386 | 383 | 395
Percentage of participants | 47.0 | 60.1 | 58.7 | 55.2
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.9775, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -8.3, 95% CI 2-sided [-16.3 to -0.2] — Adjusted Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0861, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 4.8, 95% CI 2-sided [-2.1 to 11.7] — Adjusted Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.1646, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 3.5, 95% CI 2-sided [-3.5 to 10.4] — Adjusted Difference: MK-3415A + SOC - Placebo + SOC
Statistical Analysis 4: Comparison: MK-3415 + SOC vs MK-3415A + SOC; Test type: Superiority or Other; p = 0.0025, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 11.7, 95% CI 2-sided [3.5 to 19.7] — Adjusted Difference: MK-3415A + SOC - MK-3415 + SOC
Statistical Analysis 5: Comparison: MK-6072 + SOC vs MK-3415A + SOC; Test type: Superiority or Other; p = 0.6532, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -1.4, 95% CI 2-sided [-8.3 to 5.5] — Adjusted Difference: MK-3415A + SOC - MK-6072 + SOC

3. Secondary Outcome: Percentage of Participants With CDI Recurrence in Those With Clinical Cure of the Initial CDI Episode
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive local or central lab stool test for toxigenic C. difficile following clinical cure of the initial CDI episode. Clinical cure is defined as participants who received ≤ 14 day regimen of SOC therapy and have no diarrhea (≤2 loose stools per 24 hours) for two consecutive days following completion of SOC therapy for the baseline CDI episode.
Time Frame: Up to 12 weeks
Population: Participants who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; complied with Good Clinical Practice; and achieved clinical cure of the initial CDI episode.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 169 | 299 | 286 | 327
Percentage of participants | 35.5 | 22.4 | 21.3 | 33.3
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.6505, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 1.7, 95% CI 2-sided [-6.9 to 10.7] — Adjusted Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0013, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -10.8, 95% CI 2-sided [-17.7 to -3.8] — Adjusted Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.0006, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -11.7, 95% CI 2-sided [-18.6 to -4.7] — Adjusted Difference: MK-3415A + SOC - Placebo + SOC
Statistical Analysis 4: Comparison: MK-3415 + SOC vs MK-3415A + SOC; Test type: Superiority or Other; p = 0.0007, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -13.7, 95% CI 2-sided [-22.5 to -5.2] — Adjusted Difference: MK-3415A + SOC - MK-3415 + SOC
Statistical Analysis 5: Comparison: MK-6072 + SOC vs MK-3415A + SOC; Test type: Superiority or Other; p = 0.3906, Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = -1.0, 95% CI 2-sided [-7.7 to 5.8] — Adjusted Difference: MK-3415A + SOC - MK-6072 + SOC

4. Primary Outcome: Percentage of Participants With One or More Adverse Events (AEs) During 4 Weeks Following Infusion
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended signs (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specific procedure, whether or not considered related to the medicinal product or protocol specific procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 28 days
Population: All randomized participants who received infusion of study medication, based on the treatment actually received. One participant randomized to receive MK-3415A, and two participants randomized to receive MK-6072 actually received placebo instead.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 235 | 390 | 387 | 400
Percentage of participants | 67.2 | 65.4 | 59.7 | 62.0
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.185, Miettinen and Nurminen; Percentage Difference = 5.2, 95% CI 2-sided [-2.5 to 12.8] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.323, Miettinen and Nurminen; Percentage Difference = 3.4, 95% CI 2-sided [-3.3 to 10.1] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.507, Miettinen and Nurminen; Percentage Difference = -2.3, 95% CI 2-sided [-9.1 to 4.5] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

5. Primary Outcome: Percentage of Participants With Any Drug-related AE During 4 Weeks Following Infusion
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended signs (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specific procedure, whether or not considered related to the medicinal product or protocol specific procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. A drug-related AE was an AE determined by the investigator to be related to the drug.
Time Frame: Up to 28 days
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 235 | 390 | 387 | 400
Percentage of participants | 7.2 | 8.2 | 6.2 | 5.0
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.246, Miettinen and Nurminen; Percentage Difference = 2.2, 95% CI 2-sided [-1.5 to 6.7] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.069, Miettinen and Nurminen; Percentage Difference = 3.2, 95% CI 2-sided [-0.3 to 6.8] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.464, Miettinen and Nurminen; Percentage Difference = 1.2, 95% CI 2-sided [-2.1 to 4.6] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

6. Primary Outcome: Percentage of Participants With Any Serious Adverse Events (SAEs) During 4 Weeks Following Infusion
Description: A SAE is any AE occurring at any dose or during any use of Sponsor's product that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer, or is associated with an overdose (whether accidental or intentional); or is other important medical events.
Time Frame: Up to 28 days
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 235 | 390 | 387 | 400
Percentage of participants | 27.7 | 21.5 | 14.7 | 20.0
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.027, Miettinen and Nurminen; Percentage Difference = 7.7, 95% CI 2-sided [0.9 to 14.7] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.594, Miettinen and Nurminen; Percentage Difference = 1.5, 95% CI 2-sided [-4.1 to 7.2] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.051, Miettinen and Nurminen; Percentage Difference = -5.3, 95% CI 2-sided [-10.6 to 0.0] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

7. Primary Outcome: Percentage of Participants With Any Serious Drug-related Adverse Events During 4 Weeks Following Infusion
Description: A SAE is any AE occurring at any dose or during any use of Sponsor's product that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer, or is associated with an overdose (whether accidental or intentional); or is other important medical events. A serious drug-related AE was a SAE determined by the investigator to be related to the drug.
Time Frame: Up to 28 days
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 235 | 390 | 387 | 400
Percentage of participants | 1.3 | 1.0 | 0.5 | 0.3
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.115, Miettinen and Nurminen; Percentage Difference = 1.0, 95% CI 2-sided [-0.3 to 3.5] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.170, Miettinen and Nurminen; Percentage Difference = 0.8, 95% CI 2-sided [-0.5 to 2.4] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.544, Miettinen and Nurminen; Percentage Difference = 0.3, 95% CI 2-sided [-0.9 to 1.6] — Percentage Difference: MK-3415A + SOC - Placeb + SOC

8. Primary Outcome: Percentage of Participants Who Discontinued Study Medication Due to an AE During 4 Weeks Following Infusion
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended signs (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specific procedure, whether or not considered related to the medicinal product or protocol-specific procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 28 days
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 235 | 390 | 387 | 400
Percentage of participants | 0.4 | 0.3 | 0.0 | 0.0
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.192, Miettinen and Nurminen; Percentage Difference = 0.4, 95% CI 2-sided [-0.5 to 2.4] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; p = 0.311, Miettinen and Nurminen; Percentage Difference = 0.3, 95% CI 2-sided [-0.7 to 1.4] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen; Percentage Difference = 0.0, 95% CI 2-sided [-1.0 to 1.0] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

9. Primary Outcome: Percentage of Participants With Infusion-specific AEs
Description: Infusion-specific AEs included local infusion site AEs; and systemic AEs which include nausea, vomiting, chills, fatigue, feeling hot, infusion site conditions (bruising, coldness, erythema, extravasation, pain, phlebitis, pruritus), pyrexia, arthralgia, musculoskeletal pain, myalgia, dizziness, headache, dysphonia, nasal congestion, pruritus, rash, pruritic rash, urticaria, flushing, hot flush, hypertension, and hypotension.
Time Frame: Up to 24 hours
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 235 | 390 | 387 | 400
Percentage of participants | 11.1 | 11.8 | 8.8 | 7.5
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = 3.6, 95% CI 2-sided [-1.0 to 8.7] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = 4.3, 95% CI 2-sided [0.2 to 8.5] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = 1.3, 95% CI 2-sided [-2.6 to 5.2] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

10. Secondary Outcome: Percentage of Participants ≥ 65 Years of Age at Study Entry With CDI Recurrence
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive local or central lab stool test for toxigenic C. difficile following clinical cure of the initial CDI episode.
Time Frame: Up to 12 weeks
Population: Participants ≥ 65 years of age at study entry who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 122 | 185 | 200 | 199
Percentage of participants | 26.2 | 15.1 | 17.0 | 33.2
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -6.9, 95% CI 2-sided [-16.8 to 3.5] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -18.0, 95% CI 2-sided [-26.3 to -9.6] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -16.2, 95% CI 2-sided [-24.5 to -7.7] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

11. Secondary Outcome: Percentage of Participants With a History of CDI in the 6 Months Prior to Enrollment With CDI Recurrence
Description: as for outcome 10
Time Frame: Up to 12 weeks
Population: Participants with a history of CDI in the 6 months prior to enrollment who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 69 | 103 | 96 | 109
Percentage of participants | 33.3 | 26.2 | 25.0 | 39.4
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -6.1, 95% CI 2-sided [-20.1 to 8.6] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -13.2, 95% CI 2-sided [-25.5 to -0.5] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -14.4, 95% CI 2-sided [-26.8 to -1.6] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

12. Secondary Outcome: Percentage of Participants With Clinically Severe CDI at Study Entry With CDI Recurrence
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive local or central lab stool test for toxigenic C. difficile following clinical cure of the initial CDI episode. Clinically severe CDI is defined as a Zar Score ≥ 2 based on the presence of 1 or more of the following: 1) age >60 years old (1 point); 2)body temperature >38.3°C (>100°F) (1 point); 3) albumin level ˂2.5 mg/dL (1 point); 4) peripheral white blood cell count >15,000 cells/mm^3 within 48 hours (1 point); 5) endoscopic evidence of pseudomembranous colitis (2 points); and 6) treatment in Intensive Care Unit (2 points).
Time Frame: Up to 12 weeks
Population: Participants with clinically severe CDI at study entry who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 31 | 67 | 62 | 60
Percentage of participants | 25.8 | 10.4 | 12.9 | 25.0
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = 0.8, 95% CI 2-sided [-16.9 to 21.0] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -14.6, 95% CI 2-sided [-28.3 to -1.4] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -12.1, 95% CI 2-sided [-26.2 to 1.9] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

13. Secondary Outcome: Percentage of Participants With the B1/NAP1/027 Strain of C. Difficile at Study Entry With CDI Recurrence
Description: as for outcome 10
Time Frame: Up to 12 weeks
Population: Participants with the B1/NAP1/027 strain of C. difficile at study entry who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 24 | 46 | 37 | 36
Percentage of participants | 33.3 | 26.1 | 10.8 | 36.1
Statistical Analysis 1: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -10.0, 95% CI 2-sided [-30.1 to 10.0] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -25.3, 95% CI 2-sided [-43.7 to -6.1] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

14. Secondary Outcome: Percentage of Participants With an Epidemic Strain of C. Difficile (Ribotypes 027, 014, 002, 001, 106, and 020) at Study Entry With CDI Recurrence
Description: as for outcome 10
Time Frame: Up to 12 weeks
Population: Participants with an epidemic strain of C. difficile at study entry who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 57 | 108 | 106 | 106
Percentage of participants | 24.6 | 23.1 | 19.8 | 35.8
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -11.3, 95% CI 2-sided [-24.9 to 3.9] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -12.7, 95% CI 2-sided [-24.7 to -0.5] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -16.0, 95% CI 2-sided [-27.8 to -4.0] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

15. Secondary Outcome: Percentage of Participants With Compromised Immunity at Study Entry With CDI Recurrence
Description: CDI recurrence is defined as the development of a new episode of diarrhea (3 or more loose stools in 24 or fewer hours) and a positive local or central lab stool test for toxigenic C. difficile following clinical cure of the initial CDI episode. Compromised immunity is defined as follows: an active hematological malignancy (including leukemia, lymphoma, multiple myeloma), an active malignancy requiring recent cytotoxic chemotherapy, receipt of a prior hematopoietic stem cell transplant, receipt of a prior solid organ transplant, asplenia, or neutropenia/pancytopenia due to other conditions.
Time Frame: Up to 12 weeks
Population: Participants with compromised immunity at study entry who received infusion of study medication; had a positive local stool test for toxigenic C. difficile; received protocol defined standard of care therapy within 1 day window of the infusion; and complied with Good Clinical Practice.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Number analyzed (Participants) | 55 | 87 | 78 | 92
Percentage of participants | 18.2 | 17.2 | 11.5 | 28.3
Statistical Analysis 1: Comparison: MK-3415 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -10.1, 95% CI 2-sided [-23.2 to 4.6] — Percentage Difference: MK-3415 + SOC - Placebo + SOC
Statistical Analysis 2: Comparison: MK-6072 + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -11.0, 95% CI 2-sided [-23.2 to 1.4] — Percentage Difference: MK-6072 + SOC - Placebo + SOC
Statistical Analysis 3: Comparison: MK-3415A + SOC vs Placebo + SOC; Test type: Superiority or Other; Percentage Difference = -16.7, 95% CI 2-sided [-28.4 to -4.7] — Percentage Difference: MK-3415A + SOC - Placebo + SOC

ADVERSE EVENTS:
Time Frame: Up to 90 days
Description: All randomized participants who received infusion of study medication, based on the treatment actually received. One participant randomized to receive MK-3415A, and two participants randomized to receive MK-6072 actually received placebo instead.
Groups:
- MK-3415 + SOC: Single intravenous (IV) infusion of 10 mg/kg MK-3415 + SOC for CDI
- MK-6072 + SOC: Single IV infusion of 10 mg/kg MK-6072 + SOC for CDI
- MK-3415A + SOC: Single IV infusion of 10 mg/kg MK 3415A + SOC for CDI
- Placebo + SOC: Normal saline infusion (0.9% sodium chloride) + SOC for CDI
Arm/Group | MK-3415 + SOC | MK-6072 + SOC | MK-3415A + SOC | Placebo + SOC
Serious Adverse Events (participants affected / at risk) | 104/235 | 120/390 | 94/387 | 126/400
Other Adverse Events (participants affected / at risk) | 84/235 | 116/390 | 110/387 | 103/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3415 + SOC (N=235) | MK-6072 + SOC (N=390) | MK-3415A + SOC (N=387) | Placebo + SOC (N=400)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (4) | 4 (4) | 1 (1) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 1 (1) | 3 (3) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intrapericardial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (10) | 6 (8) | 6 (7)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute graft versus host disease in intestine (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart transplant rejection (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 3 (4)
Clostridium difficile infection (Infections and infestations) | 26 (28) | 10 (13) | 18 (21) | 26 (32)
Clostridium difficile sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypopyon (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 7 (7) | 5 (5) | 11 (11)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 9 (9) | 7 (7) | 3 (3) | 11 (11)
Septic shock (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) | 4 (4)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 6 (7) | 4 (4) | 5 (5)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Zygomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perinephric collection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephritis autoimmune (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 5 (5) | 3 (3) | 6 (6)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3415 + SOC (N=235) | MK-6072 + SOC (N=390) | MK-3415A + SOC (N=387) | Placebo + SOC (N=400)
Abdominal pain (Gastrointestinal disorders) | 14 (15) | 25 (32) | 20 (21) | 24 (28)
Diarrhoea (Gastrointestinal disorders) | 18 (23) | 25 (33) | 33 (38) | 27 (42)
Nausea (Gastrointestinal disorders) | 30 (33) | 32 (38) | 33 (40) | 30 (35)
Vomiting (Gastrointestinal disorders) | 11 (13) | 23 (29) | 15 (18) | 16 (16)
Fatigue (General disorders) | 12 (13) | 7 (7) | 14 (15) | 5 (5)
Pyrexia (General disorders) | 14 (18) | 23 (26) | 13 (16) | 15 (16)
Urinary tract infection (Infections and infestations) | 15 (15) | 18 (18) | 15 (15) | 20 (21)
Headache (Nervous system disorders) | 15 (19) | 20 (23) | 22 (23) | 14 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.